CLINICAL TRIAL: NCT05436886
Title: Bioequivalence Study of Gabapentin 400 mg Capsule
Brief Title: Bioequivalence Study of Neurogabin-M (Gabapentin 400 mg) Capsule With Parketin (Gabapentin 400 mg) Capsules
Acronym: BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Merck Pvt. Ltd, Pakistan (Unknown); Center for Bioequivalence Studies and Clinical Research (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-014-GAB-2012
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers; Bioequivalence Study
Keywords: Bioequivalence Study
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Neurogabin-M 400 mg) Capsules (Experimental): A single dose consisting of one capsule of Test Drug (Neurogabin 400 mg capsule) will be administered to each of the subjects in both Periods in fasting conditions with 240 mL ambient temperature water.
  Interventions: Drug: Neurogabin (Gabapentin) 400 mg capsule; Drug: Parketin (Gabapentin) 400 mg capsule
- Reference Group (Parketin 400 mg) Capsules (Active Comparator): A single dose consisting of one capsule of Reference Drug (Parketin 400 mg capsule) will be administered to each of the subjects in both Periods under fasting conditions with 240 mL ambient temperature water.
  Interventions: Drug: Neurogabin (Gabapentin) 400 mg capsule; Drug: Parketin (Gabapentin) 400 mg capsule

INTERVENTIONS:
Drug: Neurogabin (Gabapentin) 400 mg capsule — All the subjects will receive a single dose of one capsule of either the Test Drug (Neurogabin 400 mg capsule) or Reference Drug (Parketin 400 mg capsule) in one period. if they receive Test in one period, they will alternatively receive Reference drug in the second period.
  Other Names: Gabapentin 400 mg
Drug: Parketin (Gabapentin) 400 mg capsule — All the subjects will receive a single dose of one capsule of either the Test Drug (Neurogabin 400 mg capsule) or Reference Drug (Parketin 400 mg capsule) in one period. if they receive Test in one period, they will alternatively receive Reference drug in the second period.
  Other Names: Gabapentin 400 mg

SUMMARY:
This is a single-dose, two-periods, two-sequence, two-way crossover, single oral dose bioequivalence study.

DETAILED DESCRIPTION:
This is an Open Label, Randomized, Single Dose, Two Way Cross over, Two Period, Two Treatment, Two Sequence Bioequivalence Study to compare the rate and extent of absorption of test drug Neurogabin-M 400 mg, Capsule with reference drug Parketin 400 mg Capsules in healthy adult subjects, under fasting conditions.

The study will be comprised of two Periods, I and II, each consisting of 47 hours, 11 hours before and 36 hours after the drug administration. All subjects will be divided into two groups of 12 subjects in each group. One group will be treated with the test drug (T) and the other one with reference drug (R) in Period I. After the wash-out period of 7 days, the same will receive the alternate treatment (RT) in Period II.

Blood samples at 0 hr (before drug administration) ,1.0, 1.5 , 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 14.0, 24.0, 28.0, & 36.0 hrs will be taken in both periods for quantification of drug in plasma.

All subjects will be monitored clinically for health status throughout during the periods of study and vital signs will be measured at time of check in and 1, 2, 4, 6, 8, 11, 24 and 36th hours after drug administration. ECG will be measured at time of screening in the best interest of subject safety and well being.

ELIGIBILITY:
Inclusion Criteria:

* All subjects should be healthy and free from any epidemic, contagious or measurable disease (e.g. Malaria, Dengue)
* Age range for inclusion will be 18-50 year.
* BMI for all Subjects will be between 18.5-30.0 kg/m2.
* Participant capable of understanding the informed consent.
* Non Smokers, who have not smoked in last 3 months.
* Medical history, physical examination and screening tests must fall in normal range, unless the investigator considers the abnormality to be clinically not significant.
* Clinically normal physical findings including ECG and safety laboratory values at the Screening visit and on Day -1 of each treatment period, including negative results for drugs of abuse, breath alcohol, Hepatitis B, Hepatitis C and HIV.
* Participants (who can read and understand Urdu) should be able to give informed consent, understand and sign the Informed Consent Form.
* Participants should have adequate organ function (i.e., kidney, liver and heart).
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical screening procedures and at each study period check-in.

Exclusion Criteria:

* Any active allergic disease or a history of any significant allergic disease (e.g. Rhinitis, dermatitis, asthma).
* Known hypersensitivity to Investigational drug(s).
* Abnormal results of blood and urine tests conducted at screening unless the investigator considers an abnormality to be clinically irrelevant.
* Presence or history of cardiac (e.g. Myocardial Infarction, arrythmia), renal (e.g. renal insufficiency) , hepatic (e.g. hepatic impairment) , organ insufficiency, bone marrow disease, hematological abnormality (e.g. leukemia, anemia), photosensitivity, neurological disorders) or gastrointestinal disease known to interfere with the drug absorption, distribution, metabolism or elimination (e.g. dysphagia, dyspepsia).
* History or presence of any musculo skeletal disease (e.g. Tendonitis).
* Subject donated blood (450ml) within 12 weeks minimum preceding the study.
* Alcoholic or with a history of chronic alcohol intake or consumed alcohol or Gutka in last 3 months.
* Ingestion of OTC drug, within 14 days of drug administration (e.g. aspirin, ibuprofen).
* History of intake of any prescribed medicine (e.g. Captopril, Sumatriptan) during a period of 30 days, prior to drug administration day of study.
* Ingestion of investigational drug within 30 days, prior to investigational drug administration in the study.
* Ingestion of any known hepatic or renal clearance altering agents (e.g. erythromycin, cimetidine, barbiturates, phenothiazines, etc.) for a period of 30 days, prior to study initiation. Drug interaction section at 5.10 and Warnings section at 5.11 should be considered.
* Subjects with an uncontrolled medical condition (i.e., hypertension, cardiac arrhythmias, CHF) that places the patient at risk by participating in the study.
* Subjects with known HIV, hepatitis B or C infection or autoimmune diseases.
* History of drug exposure which, in the opinion of Investigator, amounts to drug abuse (e.g. Amphetamine).
* Participation in other drug studies within three months prior to study initiation.
* Subjects who is unable to or likely to be non-compliant with protocol requirements or restrictions.
* Limited mental capacity to the extent that the subject is unable to provide legal consent and information regarding the side effects or tolerance of the study drug.
* Pregnancy or breast feeding, women of child bearing age who are not using a recognized form of contraception for at least last 30 days or using hormonal contraception, are also excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2013-07-05 (Actual); Study Completion 2013-09-10 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-36 hours post dose
  Maximum plasma concentration of Gabapentin
AUC last (AUC 0-t) | 0-36 hours post dose
  Area under plasma concentration time curve from zero to time of the last measurable concentration
AUC total (AUC 0-∞) | 0-36 hours post dose
  Area under the plasma concentration-time curve from zero to infinity.

SECONDARY OUTCOMES:
Tmax | 0-36 hours post dose
  Time to reach maximum drug concentration in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad R Shah, PhD, Principal Investigator — Center for bio-equivalence, and clinical research, university of karachi; Dr. Naghma Hashmi (Co-PI), PhD, Principal Investigator — Center for bio-equivalence, and clinical research, university of karachi
Locations (1):
- Center for Bioequivalence Studies and clinical research (CBSCR), ICCBS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No